CLINICAL TRIAL: NCT02214966
Title: Influence of Food on the Bioavailability of 80 mg Telmisartan / 10 mg Ramipril Fixed Dose Combination in Healthy Male and Female Volunteers (an Open-label, Randomised, Single-dose, Two-sequence, Two-period Crossover Study)
Brief Title: Influence of Food on the Bioavailability of Telmisartan / Ramipril Fixed Dose Combination in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1236.3
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; Ramipril

ARMS (2):
- Telmisartan/Ramipril, fed (Experimental)
  Interventions: Drug: Telmisartan/Ramipril, fixed dose combination tablet; Other: high fat, high caloric meal
- Telmisartan/Ramipril, fasted (Active Comparator)
  Interventions: Drug: Telmisartan/Ramipril, fixed dose combination tablet

INTERVENTIONS:
Drug: Telmisartan/Ramipril, fixed dose combination tablet
Other: high fat, high caloric meal
  Arms: Telmisartan/Ramipril, fed

SUMMARY:
The objective was to investigate the relative bioavailability of the fixed dose combination (FDC) tablet (80 mg telmisartan / 10 mg ramipril) after food intake in comparison to the bioavailability of the FDC tablet while fasting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age ≥18 and ≤55 years
* Body mass index (BMI) ≥18.5 and ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* Inability to refrain from smoking during 24 hours prior to dosing and 24 hours after dosing
* Alcohol abuse (more than 60 g/day) or inability to stop alcoholic beverages for 24 hours prior to dosing and up to the last sampling time point
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration of trial drug or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g. repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hyperkalemia, hypokalemia, family history of Long QT Syndrome)
* Any history of relevant low BP
* Supine blood pressure at screening of systolic <110 mm Hg and diastolic <60 mm Hg
* History of urticaria
* History of angioneurotic edema
* Hereditary fructose intolerance
* Salt and/or volume depletion

For female subjects:

* Pregnancy / positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion
* No adequate contraception during the study and until 1 month of study completion, i.e. implants, injectables, combined oral contraceptives, intrauterine device, sexual abstinence (for at least 1 month prior to enrolment), vasectomised partner (vasectomy performed at least 1 year prior to enrolment) or surgical sterilisation (incl. hysterectomy). Females, who have not a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide)
* Currently lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2007-10; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analytes in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours after drug administration
AUC0-24 (area under the concentration-time curve of the analytes in plasma over one dosing interval from 0 to 24h) | up to 96 hours after drug administration
Cmax (maximum measured concentration of the analytes in plasma) | up to 96 hours after drug administration
AUC0-tz (area under the concentration-time curve of ramipril in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 96 hours after drug administration
tmax (time from dosing to the maximum concentration of the analytes in plasma) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
λz (terminal rate constant in plasma) | up to 96 hours after drug administration
t1/2 (terminal half-life of the three analytes in plasma) | up to 96 hours after drug administration
MRTpo (mean residence time of the analytes in the body after po administration) | up to 96 hours after drug administration
CL/F (apparent clearance of the analytes in the plasma after extravascular administration) | up to 96 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 96 hours after drug administration
Number of patients with adverse events | up to 54 days
Assessment of tolerability by investigator on a 4-point scale | Day 5 of each treatment period
Number of patients with clinically significant changes in Vital Signs (Blood Pressure, Pulse Rate) | up to 54 days
Number of patients with clinically significant changes in laboratory tests | up to 54 days
Number of patients with clinically significant changes in Electrocardiogram (ECG) | up to 54 days
AUC0-tz (area under the concentration-time curve of ramiprilat and telmisartan in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 96 hours after drug administration